CLINICAL TRIAL: NCT02670564
Title: Allogeneic Stem Cell Transplant for Children and Adolescents With Acute Lymoblastic Leukemia FORUM - Pharmacogenomic Study (add-on Study)
Brief Title: ALL SCTped FORUM - Pharmacogenomic Study (add-on Study)
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Swiss Pediatric Oncology Group (Other)
Collaborators: ALL SCTped Forum (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: ZH 2014-0535; NZ 2015-069 (Registry Identifier: Commission compétente); GE 15-034 (Registry Identifier: Commission compétente)
Record Dates: First submitted 2015-07-03; First posted 2016-02-02 (Estimated); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Acute Lymphoblastic Leukemia
Keywords: pharmacogenetics; busulfan; treosulfan; hematopoietic stem cell transplantation; fludarabine; pediatric patients; TBI; leukemia; leukemia, lymphoid; precursor cell lymphoblastic Leukemia-Lymphoma; Immune System disease; Immunoproliferative Disorders; stem cell transplantation; children and adolescent; high risk acute lymphoblastic leukemia; NCT01949129 add-on; ALL SCTped FORUM
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia; Leukemia, Lymphoid; Immune System Diseases; Immunoproliferative Disorders | interventions — Pharmacogenomic Testing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Total body irradiation (TBI) (Experimental): The Pharmacogenomics add-on requires 2X 5ml blood EDTA for further DNA analyses.
  Note this is an add-on study to NCT 01949129, THE ALL SCTped FORUM study. Please refer to the main study for further details.
  Interventions: Genetic: Pharmacogenomics
- Busulfan (Experimental): The Pharmacogenomics add-on requires 2X 5ml blood EDTA for further DNA analyses.
  Note this is an add-on study to NCT 01949129, THE ALL SCTped FORUM study. Please refer to the main study for further details.
  Interventions: Genetic: Pharmacogenomics; Other: Busulfan plasma level measurements
- Treosulfan (Experimental): The Pharmacogenomics add-on requires 2X 5ml blood EDTA for further DNA analyses.
  Note this is an add-on study to NCT 01949129, THE ALL SCTped FORUM study. Please refer to the main study for further details.
  Interventions: Genetic: Pharmacogenomics

INTERVENTIONS:
Genetic: Pharmacogenomics — Blood samples (2x5ml EDTA tubes) should be collected just before the start of the conditioning regimen from every patient regardless of therapeutic arm by every centre and stored ≤-20°C Patient should be in remission (MRD negative) for this sampling, otherwise the sample should be taken using a mouth swab/saliva (not intravenously).
  For second transplant patients, please provide DNA taken before first transplant or a fresh saliva samples.
  Other Names: DNA analyses
Other: Busulfan plasma level measurements — Bu PK analysis after the first dose of IV Bu (+potential subsequent ones).
  Blood sampling:
  ->For Bu 4 X/d: Before the first Bu dose (Time 0), then straight after the end of infusion (Time 1), then at 15 min (Time 2), 30 min (Time 3), 1 hour (Time 4) and 4 hour (Time 5) after the end of infusion
  ->For Bu 1 X/d: Before the first Bu dose (Time 0), then straight after the end of infusion (Time 1), then at 1 hour (Time 2), 3 hour (Time 3), 5 hour (Time 4), 7 hour (Time 5) and 11 hour (Time 6) after the end of infusion.
  For centers not performing BU TDM, perform Dried Blood Sampling (DBS) analysis:
  -> 0.5ml blood sample should be collected and 5µl spotted onto DBS cards in duplicate. Dry them max 5 hours and then keep in a sealed envelope and store at -80°C, as below
  Arms: Busulfan

SUMMARY:
Pharmacogenomics (PG) offers the opportunity to individualize treatment according to patient genetic variations which influence activity of enzyme metabolizing or acting in the pathway of prescribed chemotherapy drugs.

This add-on research aims to prospectively investigate variations in several candidate genes related to all types of chemotherapeutic drugs and TBI used in the main related study NCT 01949129, THE ALL SCTped FORUM study for their potential role as predictive biomarkers of PK variability and outcome of myeloablative therapy for pediatric patients receiving an allogeneic hematopoietic stem cell transplantation in acute lymphoblastic leukemia.

DETAILED DESCRIPTION:
Note this is an add-on study to NCT 01949129, THE ALL SCTped FORUM study. Please refer to the main study for further details.

Busulfan (Bu) is a key compound in conditioning myeloablative regimens for patients undergoing hematopoietic stem cell transplantation (HSCT). Bu has been long used for the treatment of patients with leukemia and some congenital disorders; advantages and disadvantages of such treatment are well described. However, although Bu treatment has been shown to be effective, its use may be limited by related adverse events such as veno-occlusive disease (VOD), interstitial pneumonitis, acute Graft vs Host Disease (GVHD), and seizures. Thus, novel therapies are being investigated as well as the pharmacogenetics of these drugs. One of alternative drugs that may replace Bu due to its lower toxicity profile is Treosulfan (Treo). Fludarabine (Flu) is usually used in combination with Bu or Treo as an alternative to cyclophosphamide (Cy) also due to its lower toxicity. Thus, the Bu/Flu regimen is now being used more often than the previously more common Bu/Cy regimen. However, improvement to the regimen is still needed for reducing adverse drug effects. Pharmacogenomics (PG) offers the opportunity to individualize treatment according to patient genetic variations which influence activity of enzyme metabolizing or acting in the pathway of prescribed chemotherapy drugs.

This add-on research aims to prospectively investigate variations in several candidate genes (e.g GST, DCK and DNA repair pathway genes) related to all types of chemotherapeutic drugs (Bu/Flu/Thio; Treo/Flu/Thio and TBI/VP16) used in this protocol for their potential role as predictive biomarkers of pharmacokinetics (PK) variability and outcome of myeloablative therapy for pediatric patients receiving an allogeneic HSCT in acute lymphoblastic leukemia

For the busulfan arm countries: a cross-validation of busulfan quantification is performed. All Bu Therapeutic Drug Monitoring participating at the main ALL SCTped FORUM study will be assessed for the accuracy (%) and trueness (%) of 8 blinded Bu Quality Control samples. Criteria of acceptance are set according to FDA and ICH guidelines.

Blood samples will be collected prior to initiation of therapy for DNA banking and DNA analysis (for all patients), for DNA analysis (TBI/VP16, Bu/Flu/Thiotepa and Treo/Flu/Thiotepa groups) and PK analysis (only for the Bu group). PK and pharmacogenomic data will then be correlated with the studied outcomes (e.g.Veno-occlusive disease, Graft vs host disease, Treatment Related Mortality, Events Free Survival, Overall Survival).

Recruitment:

Patients (children) age 0-18 will be recruited in each arm. No oral Bu is allowed in this study.

Shipment (when there is a minimum of 10 patients) Send all the materials listed to: Dr Marc Ansari, Plateforme d'Hématologie et Oncologie Pédiatrique (CANSEARCH research laboratory), Faculté de Médecine, Bâtiment Tulipe, 5th floor, Av De La Roseraie 64, GENEVE 1205 Switzerland.

Contact Dr. Ansari's laboratory prior to shipment: Phone (+41 79 55 36 100) and e-mail (research@cansearch.ch). All shipments must be sent frozen by a carrier guaranteeing overnight delivery with the indication "Pharmacogenomic study" on the face of the parcel.

ELIGIBILITY:
Note this is an add-on study to NCT 01949129, THE ALL SCTped FORUM study. Please refer to the main study for further details.

Gender

* Both: both female and male participants are being studied

Age Limits

* Minimum Age: N/A
* Maximum Age: age at time of screening less than 18 years old

Accepts Healthy Volunteers: no

Eligibility Criteria

Inclusion Criteria:

* Patients with ALL (except for patients with B-ALL)
* indication for allogeneic HSCT
* complete remission (CR) before HSCT
* written consent of the parents (legal guardian) and, if necessary, the minor patient via "Informed Consent Form"
* no pregnancy
* no secondary malignancy
* no previous HSCT
* HSCT is performed in a study participating centre

Exclusion Criteria:

* Non Hodgkin-Lymphoma
* ALL with extramedullary involvement with indication for TBI
* CNS involvement at the timepoint of screening
* Trisomy 21
* The whole protocol or essential parts are declined either by patient himself/herself or the respective legal guardian
* No consent is given for saving and propagation of anonymous medical data for study reasons
* Severe concomitant disease that does not allow treatment according to the protocol at the investigator's discretion (e.g. malformation syndromes, cardiac malformations, metabolic disorders)
* Karnofsky / Lansky score < 50%
* Subjects unwilling or unable to comply with the study procedures

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1000 (Estimated)
Dates: Start 2013-04; Primary Completion 2021-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Genetic variants in participants as a marker of risk of Adverse events and/or Efficacy of the studied agents | through study completion, an average of 2 years
  Genotyping of candidates genes related to pharmacokinetics and pharmacodynamics of the studied agents.
  Association study between the herein genetic variants and the below mentioned phenotypes (odd ratio).

SECONDARY OUTCOMES:
Number of participants with acute Graft-versus-host disease (aGvHD) according to the Glucksberg scale and Seattle criteria | 18 months after inclusion of first patient, afterwards, annually up to 10 years
Number of participants with chronic Graft-versus-host disease (cGvHD) according to the Glucksberg scale and Seattle criteria | 18 months after inclusion of first patient, afterwards, annually up to 10 years
Number of participants with VOD/SOS according to the Seattle criteria | 18 months after inclusion of first patient, afterwards, annually up to 10 years
Number of participants with Neutrophil recovery as a measure of Safety and Tolerability | 18 months after inclusion of first patient, afterwards, annually up to 10 years
  defined as the first of 3 consecutive days with an absolute neutrophil count of 0.5x10^9/L or higher
Number of participants with Platelet recovery as a measure of Safety and Tolerability | 18 months after inclusion of first patient, afterwards, annually up to 10 years
  Defined as the first of 3 consecutive days with platelet counts higher that 20x10^9/L without transfusion
Number of participants with Primary graft failure or rejection as a measure of Safety and Tolerability | 18 months after inclusion of first patient, afterwards, annually up to 10 years
  Defined by persistent pancytopenia with no evidence of hematologic recovery of donor cells beyond 28 days after transplantation, and secondary graft failure by a rapid decrease in neutrophil count after successful engraftment
Transplant related mortality (TRM) | 18 months after inclusion of first patient, afterwards, annually up to 10 years
  the time of transplant until all causes of death after transplant not related to relapse
Event free survival (EFS) | 18 months after inclusion of first patient, afterwards, annually up to 10 years
  the time of transplant until death, relapse or graft failure, whichever occurs first.
Overall survival (OS) | 18 months after inclusion of first patient, afterwards, annually up to 10 years
  the time between transplantation and death due to any causes
Cumulative incidence of relapse | 18 months after inclusion of first patient, afterwards, annually up to 10 years

OTHER OUTCOMES:
Administered Bu dose(mg) per day | Measures assessed at time of conditioning (up to 5days)
  Bu pharmacokinetics profile
Target Bu plasma concentration(ng/ml) | Measures assessed at time of conditioning (up to 5days)
  Bu pharmacokinetics profile
Target Bu Area under the plasma concentration versus time curve (AUC) (min*ng/ml) | Measures assessed at time of conditioning (up to 5days)
  Bu pharmacokinetics profile
Measured Area under the plasma concentration versus time curve (AUC) of Bu (min*ng/ml) | Measures assessed at time of conditioning (up to 5days)
  Bu pharmacokinetics profile
Measured maximum plasma Bu concentration (Cmax, ng/ml) | Measures assessed at time of conditioning (up to 5days)
  Bu pharmacokinetics profile
Measured minimum plasma Bu concentration (Cmin, ng/ml) | Measures assessed at time of conditioning (up to 5days)
  Bu pharmacokinetics profile
Measured steady state plasma Bu concentration (Css, ng/ml) | Measures assessed at time of conditioning (up to 5days)
  Bu pharmacokinetics profile
Measured Clearance of Bu (ml/min/kg) | Measures assessed at time of conditioning (up to 5days)
  Bu pharmacokinetics profile

CONTACTS AND LOCATIONS:
Overall Officials: Christina Peters, Prof. MD PhD, Study Chair — St. Anna Kinderspital, Vienna, Austria; Peter Bader, Prof. MD PhD, Study Chair — Klinik für Kinder- u. Jugendheilkunde III, Johann Wolfgang Goethe Universität, Frankfurt, Germany; Franco Locatelli, Prof. MD PhD, Study Chair — Department of Pediatric Hematology and Oncology IRCCS Ospedale, Rome, Italy; Marc Ansari, MD, PD, Principal Investigator — Département de Pédiatrie, Hôpital Cantonal de Genève
Locations (4):
- Switzerland (4):
  - Hôpital Cantonal de Genève, Département de Pédiatrie, Geneva, Cansearch Laboratory
  - Universitäts-Kinderspital beider Basel (UKBB), Onkologie/Hämatologie, Basel
  - HUG Hôpitaux Universitaire de Genève, Unité d'onco-hématologie pédiatrique, Geneva
  - Universitäts-Kinderspital, Zurich

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Cansearch laboratory — https://cansearch.ch/en/
- See also: St. Anna Kinderkrebsforschung — http://www.kinderkrebsforschung.at/